CLINICAL TRIAL: NCT05675072
Title: A Phase II/III,Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of FB2001 for Inhalation in Patients With Mild to Moderate COVID-19
Brief Title: Evaluate the Efficacy and Safety of FB2001 for Inhalation in Patients With Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB2001-302
Record Dates: First submitted 2023-01-02; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Mild to Moderate COVID-19
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); FB2001; Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — FB2001; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB2001 group (Experimental): FB2001 will be administered by nebulized inhalation, plus Standard Of Care(SOC)
  Interventions: Drug: FB2001
- Placebo group (Placebo Comparator): Placebo will be administered by nebulized inhalation, plus Standard Of Care(SOC)
  Interventions: Drug: FB2001 placebo

INTERVENTIONS:
Drug: FB2001 — FB2001 for Inhalation will be reconstituted with normal saline prior to nebulized inhalation. FB2001 will be administered by nebulized inhalation.
  Other Names: FB2001 for Inhalation
  Arms: FB2001 group
Drug: FB2001 placebo — FB2001 placebo will be reconstituted with normal saline prior to nebulized inhalation. FB2001 placebo will be administered by nebulized inhalation.
  Other Names: placebo
  Arms: Placebo group

SUMMARY:
This study is a double-blind,randomized,placebo-controlled study to evaluate the efficacy and safety of FB2001 for Inhalation in patients with mild to moderate Coronavirus Disease 2019(COVID-19). A total of about 1336 subjects are planned to be enrolled. The subjects will be randomized in a 1:1 ratio to FB2001 group or placebo group while both receiving standard of care treatment.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID -19) is a respiratory illness that can spread from person to person. The infectious agent that causes COVID -19 is a novel coronavirus, named severe acute respiratory syndrome coronavirus 2(SARS-CoV-2), was first identified during a recent outbreak in December 2019, Patients with COVID-19 have symptoms of fever, cough, and shortness of breath along with non-specific symptoms including myalgia and fatigue.

FB2001 is a small-molecule inhibitor of coronavirus 3CL protease(3CLpro). In phase I clinical trial, FB2001 for Inhalation were safe and tolerable well in healthy subjects, and were projected to be effective in patients according to its pharmacokinetic profile.

This study is a double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of FB2001 for Inhalation in patients with mild to moderate Coronavirus Disease 2019 (COVID-19). The subjects will be randomized in a 1:1 ratio to FB2001 group or placebo group while both receiving standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female;
* Confirmed SARS-CoV-2 infection as determined by Reverse Transcription - Polymerase Chain Reaction(RT -PCR) in any specimen collected within 5 days prior to randomization.

Note: RT-PCR is the preferred method; however, with evolving approaches to laboratory confirmation of SARS-CoV-2 infection, other molecular or antigen tests that detect viral RNA or protein are allowed if authorized for use in the country;

* Patients with mild or moderate COVID-19.
* Initial onset of signs/symptoms attributable to COVID -19 within 3 days prior to the day of randomization and at least one of the specified signs/symptoms attributable to COVID -19 present on the day of randomization;
* Women of childbearing potential who have a negative serum or urine pregnancy test prior to the first study dose;
* Patient who is willing to cooperate and able to participate in the trial, adhered to all requirements of the protocol, and provided written informed consent.

Exclusion Criteria:

* Patients who are currently or are expected to potentially progress to severe/critical COVID-19 within 48 h of randomization;
* Patients with chronic respiratory diseases, including bronchial asthma and chronic obstructive pulmonary disease etc.
* Known history of moderate-severe liver impairment (e.g., Child-Pugh grade B or C, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5x upper limit normal (ULN) , or acute liver failure within 6 months prior to screening;.
* Known history of severe renal impairment (e.g., Chronic Kidney Disease-Improved Prediction Equations(CKD-EPI)formula based on serum creatinine, estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2), or was receiving renal replacement therapy, such as peritoneal dialysis or hemodialysis, within 6 months prior to screening;
* Impaired immune system (including patients treated with systemic corticosteroids or other immunosuppressive agents, or cancer progression or recurrence)
* Suspected or confirmed concurrent active systemic infections other than COVID-19 that may interfere with the assessment of response to study interventions.
* Need for radiotherapy, chemotherapy, emergency surgery or surgical treatment at screening, or other emergencies (e.g. acute coronary syndrome, acute pulmonary embolism, etc.).
* Patients with a history of cardiopulmonary resuscitation or major surgery within 30 days prior to randomization, and patients with other potentially life-threatening clinical conditions or other emergencies.
* History of hypersensitivity or other contraindications to any component of the study intervention.
* Patients who received or expected to receive anti-SARS-CoV-2 viral drugs (e.g., nirmatrelvir/ritonavir, molnupiravir, etc.) within 14 days prior to randomization.
* Have received (within 30 days prior to randomization or within 5 half-lives, whichever is longer) or expect to receive COVID-19 monoclonal antibody or recovery COVID-19 plasma therapy.
* Any SARS-CoV-2 vaccination within 3 months prior to randomization.
* Within 28 days or 5 half-lives (whichever is longer) prior to randomization or in clinical studies with other investigational drugs or devices, including studies for COVID-19.
* Mental illnesses that, in the judgment of the investigator, are not appropriate for participation in this study.
* Any other situation that the investigator believes may affect the subject's informed consent or adherence to the protocol, or the subject's participation in the study may affect the outcome of the study or his or her own safety, in the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1336 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to sustained recovery of COVID-19-related signs/symptoms | Up to Day 29
  Sustained recovery of a COVID-19-related sign/symptom is defined as a COVID-19-related sign/symptom score of 0 for 3 consecutive days, i.e., disappearance of COVID-19-related symptoms or return to the status prior to the onset of COVID-19.

SECONDARY OUTCOMES:
Proportion of participants who have progression of COVID-19 . | Up to Day 29
  Disease progression is defined as disease severity from mild to moderate or severe or critical, or moderate to severe or critical, or all-cause death
Time to sustained alleviation of COVID-19-related sign/symptom. | Up to Day 29
  Sustained alleviation of COVID-19-related signs/symptoms are defined as the COVID-19-related sign/symptom score from 0 or 1 to 0 at baseline or from 2 or 3 to 1 or 0 at baseline for 3 consecutive days.
Time to sustained recovery of 5 key COVID-19-related sign/symptom | Up to Day 29
  Sustained recovery of a COVID-19-related sign/symptom is defined as a COVID-19-related sign/symptom score of 0 for 3 consecutive days, i.e., disappearance of COVID-19-related symptoms or return to the status prior to the onset of COVID-19.
Time to sustained alleviation of 5 key COVID-19-related sign/symptom | Up to Day 29
  Sustained alleviation of COVID-19-related signs/symptoms are defined as the COVID-19-related sign/symptom score from 0 or 1 to 0 at baseline or from 2 or 3 to 1 or 0 at baseline for 3 consecutive days.
Proportion of participants who experience sustained recovery of COVID-19 sign/symptom | Day 3 to Day 21
  no special description
Proportion of participants who experience sustained alleviation of COVID-19-related sign/symptom | Day 3 to Day 21
  no special description
Duration of each targeted COVID-19-related sign/symptom. | Up to Day 29
  no special description
Time to sustained virus clearance of SARS-CoV-2 in nasopharyngeal swabs | Up to Day 29
  no special description
Changes in SARS-CoV-2 viral load | Up to Day 29
  no special description
Change in EQ-5D-5L index score | Up to Day 29
  The Euroquol Quality of Life 5-Dimension 5-Level Scale(EQ-5D-5L) index score consists of five dimensions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each dimension has five scales: no difficulty, a little difficulty, moderate difficulty, severe difficulty, and very severe difficulty

OTHER OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events(TEAEs) | Up to Day 29
  safety evaluation
Incidence of withdrawals due to Adverse Events(AEs) | Up to Day 29
  safety evaluation
Incidence of Serious Adverse Events(SAEs) | Up to Day 29
  safety evaluation
Safety as determined by abnormality in haematology | Up to Day 29
  Measurement of white blood cell (WBC) count, red blood cell (RBC) count, haemoglobin (Hb), neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, Platelets absolute count.
Safety as determined by abnormality in clinical chemistry | Up to Day 29
  Measurement of sodium, potassium, urea/blood urea nitrogen (BUN), creatinine, albumin, calcium, phosphate, glucose, c-reactive protein (CRP), alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transpeptidase (GGT), total bilirubin, conjugated bilirubin, creatine kinase.
Incidence of treatment-related grade 3 or above TEAEs | Up to Day 29
  safety evaluation
Safety as determined by abnormality in urinalysis | Up to Day 29
  Measurement of glucose, protein, blood and microscopy.
Safety as determined by abnormality in Coagulation. | Up to Day 29
  Measurement of international normalised ratio (INR), prothrombin time, activated partial thrombin time (aPTT).
Incidence of treatment-related adverse events (TRAEs) | Up to Day 29
  safety evaluation
Incidence of discontinuation of study treatment due to TEAEs | Up to Day 29
  safety evaluation
Incidence of abnormal 12-lead electrocardiogram (ECG) | Up to Day 29
  Results for P wave PR interval, QRS duration, QT interval, QTcF interval, RR interval, and heart rate will be analyzed.
Safety as determined by abnormal vital signs (blood pressure, pulse rate, body temperature, and respiratory rate) | Up to Day 29
  Measurement of systolic blood pressure (mm Hg), diastolic blood pressure (mm Hg), pulse rate (beats per minute), body temperature (in degree Celsius), respiratory rate (breaths per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, Study Director — Frontier Biotechnologies Inc.
Locations (1):
- Shenzhen Third People's Hospital, Shenzhen, Guangdong, China